CLINICAL TRIAL: NCT07050589
Title: A Community-Based Recreation Program to Improve Function and Quality of Life in Older Adults
Brief Title: Group Recreation to Enhance Function Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Nikhil Satchidanand, Assistant Professor of Internal Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00008757
Record Dates: First submitted 2025-04-08; First posted 2025-07-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Physical Functioning; Cognitive Functioning
Keywords: walking; balance; strength; attention; memory; interference inhibition; dual-task; artmaking; exergaming
MeSH Terms: interventions — Exercise; Reproductive Techniques, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program (Experimental): Program participants will receive the recreation-based program.
  Interventions: Behavioral: Exercise and art
- Control (No Intervention): Control participants will receive no recreation-based program.

INTERVENTIONS:
Behavioral: Exercise and art — Weekly SMARTfit dual-task exergaming and group art-making
  Arms: Program

SUMMARY:
Investigators will develop and deliver a community-based recreation program, delivering group artmaking and group SMARTfit dual-task exergaming to community-dwelling older adults. The program will be delivered through the Buffalo-Niagara YMCA. Outcomes of interest are change in cognitive function and change in physical functioning, inresponse to 24 weeks of weekly training.

ELIGIBILITY:
Inclusion Criteria

* > = 60 years of age
* have no more than MCI (MoCA score ≥ 24 points)
* have no contraindications to exercise, guided by the American College of Sports Medicine
* fluent in English

Exclusion Criteria

* have a condition that would prevent safe participation in the exercise, as determined by the Physical Activity Readiness Questionnaire for Older Adults (PAR-OA);
* have severe neurological disease
* have severe psychiatric illness
* have a likelihood of withdrawing from the study due to severe illness or a life expectancy of < 6 mo
* have experienced a lower or upper limb amputation
* have greater than mild cognitive impairment (MoCA score < 24 points).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function: Attention | From enrollment to week 8 and then week 16
  Change in performance on the Trail-Making Test

SECONDARY OUTCOMES:
Balance | From enrollment to week 8 and then week 16
  Change in balance assessed by the Four Stage Balance Test
Dual-Task Performance | From enrollment to week 8 and then week 16
  Dual task performance assessed using the Timed Up and Go-Dual Task
Cognitive Function: Interference Inhibition | baseline to week 8, through week 16
  Change in performance on the Stroop Test

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo-Niagara YMCA, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests to access deidentified participant data can be submitted starting 12 months after article publication and the data will be made accessible for up to 12 months. Access to IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, contact NS1@buffalo.edu.
Supporting Information: Study Protocol
Time Frame: 06/15/2026 - 05/14/2027
Access Criteria: Access to IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).